CLINICAL TRIAL: NCT00802282
Title: Effects of Psilocybin and Spiritual Practice on Persisting Changes in Attitudes and Behavior
Brief Title: Psilocybin and Spiritual Practice
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Fetzer Institute (Other); The CSP Fund of the San Francisco Foundation (Unknown)
Responsible Party: Principal Investigator, Roland Griffiths, Professor, Department of Psychiatry, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NA_00020767
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: healthy volunteers; spirituality; psilocybin; meditation
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): First of 5 groups, as described in the protocol and to which volunteers are blinded
  Interventions: Drug: psilocybin; Behavioral: Intensity of support for spiritual practice; Behavioral: Number of sessions
- 2 (Experimental): Second of 5 groups, as described in the protocol and to which volunteers are blinded
  Interventions: Drug: psilocybin; Behavioral: Intensity of support for spiritual practice; Behavioral: Number of sessions
- 3 (Experimental): Third of 5 groups, as described in the protocol and to which volunteers are blinded
  Interventions: Drug: psilocybin; Behavioral: Intensity of support for spiritual practice; Behavioral: Number of sessions
- 4 (Experimental): Fourth of 5 groups, as described in the protocol and to which volunteers are blinded
  Interventions: Drug: psilocybin; Behavioral: Intensity of support for spiritual practice; Behavioral: Number of sessions
- 5 (Experimental): Fifth of 5 groups as described in the protocol and to which volunteers are blinded
  Interventions: Drug: psilocybin; Behavioral: Intensity of support for spiritual practice; Behavioral: Number of sessions

INTERVENTIONS:
Drug: psilocybin — dose manipulation as described in the protocol and to which volunteers are blinded
Behavioral: Intensity of support for spiritual practice — Volunteers will be assigned to standard or high support, as described in the protocol
Behavioral: Number of sessions — Volunteers will be assigned to either 2 or 3 sessions, as described in the protocol

SUMMARY:
This study will investigate the effects of psilocybin dose and the frequency and intensity of support activities for spiritual practice (e.g., meditation) on a battery of attitudinal and behavioral outcome measures in 75 healthy volunteers who are interested in pursuing a program of spiritual practices with the intention applying spiritual insights and knowledge to everyday life. After screening and study enrollment, each volunteer will be assigned to one of five groups that vary in dose, frequency and intensity of support for spiritual practice, and number of psilocybin sessions (either 2 or 3 sessions). The psilocybin dose manipulation will be double-blind. Volunteers will be told that in each of sessions 1, 2, and 3, he/she could receive a very low, low, moderate, moderately high, or high dose of psilocybin. They will be told that each participant will receive 2 or more dose levels of psilocybin over the 2 or 3 sessions, and all participants will have one or more sessions in which he or she receives a moderately high or high dose of psilocybin. The duration of each volunteer's participation will be approximately 6 to 8 months. Each volunteer will receive several hours of preparation with the study guides in the month prior to the first psilocybin session; the first two sessions will be separated by one month. Various measures will be assessed before, during and immediately after sessions. A battery of longitudinal measures will be evaluated immediately after study enrollment, 3 weeks after the second psilocybin session, and 4 months after the second psilocybin session (6 months after study enrollment). For purposes of controlling expectancies through the 6 month follow-up evaluation, volunteers and guides will not know which volunteers or how many volunteers will be scheduled for a third session.

ELIGIBILITY:
Eligibility criteria for volunteers who will receive psilocybin

Inclusion Criteria:

* 21 to 70 years old
* Have given written informed consent
* Have a high school level of education
* Be healthy and psychologically stable as determined by screening for medical and psychiatric problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests.
* Have an active interest in exploring and developing their spiritual lives
* Cigarette smokers must agree to abstain from smoking on psilocybin session days from 1 hour before psilocybin administration until at least 6 hours after psilocybin administration.
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the volunteer does not routinely consume caffeinated beverages, he or she must agree not to do so on session days.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of each psilocybin administration. Exceptions include caffeine and nicotine.
* Agree not to take any PRN medications on the mornings of psilocybin sessions
* Agree that for one week before each psilocybin session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.

Exclusion Criteria:

General medical exclusion criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), or TIA in the past year
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting pharmacological effect on serotonin neurons or medications that are MAO inhibitors. For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* More than 20% outside the upper or lower range of ideal body weight

Psychiatric Exclusion Criteria:

* Current or past history of meeting DSM-IV criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder.
* Current or past history within the last 5 years of meeting DSM-IV criteria for alcohol or drug dependence (excluding caffeine and nicotine) or severe major depression.
* Have a first or second degree relative with Schizophrenia, Psychotic Disorder (unless substance induced or due to a medical condition), or Bipolar I or II Disorder.
* Currently meets DSM-IV criteria for Anorexia Nervosa, Bulimia Nervosa, or other psychiatric conditions judged to be incompatible with establishment of rapport or safe exposure to psilocybin

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-08; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Hood Mysticism Scale | At end of sessions
States of Consciousness Questionnaire | At end of sessions
Persisting Effects Questionnaire | 3 weeks after each session

SECONDARY OUTCOMES:
Daily spiritual experiences scale | Baseline, 3 weeks after second session, 6 months, and 3 weeks after the third session
A battery assessing various measures of gratitude, forgiveness, religious coping, death attitude, life purpose, life satisfaction, and psychological functioning | Baseline, 3 weeks after second session, 6 months, and 3 weeks after the third session
Blood markers of stress and immune function | Baseline, 3 weeks after second session, 6 months, and 3 weeks after the third session
Brief symptom inventory | Baseline, one week after each session, and at 6 months
Visual effects questionnaire | Baseline, 6 months, and 3 weeks after the third session

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Griffiths, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Griffiths RR, Richards WA, McCann U, Jesse R. Psilocybin can occasion mystical-type experiences having substantial and sustained personal meaning and spiritual significance. Psychopharmacology (Berl). 2006 Aug;187(3):268-83; discussion 284-92. doi: 10.1007/s00213-006-0457-5. Epub 2006 Jul 7. PMID 16826400
- [Background] Griffiths R, Richards W, Johnson M, McCann U, Jesse R. Mystical-type experiences occasioned by psilocybin mediate the attribution of personal meaning and spiritual significance 14 months later. J Psychopharmacol. 2008 Aug;22(6):621-32. doi: 10.1177/0269881108094300. Epub 2008 Jul 1. PMID 18593735
- [Background] Johnson M, Richards W, Griffiths R. Human hallucinogen research: guidelines for safety. J Psychopharmacol. 2008 Aug;22(6):603-20. doi: 10.1177/0269881108093587. Epub 2008 Jul 1. PMID 18593734
- [Derived] Griffiths RR, Johnson MW, Richards WA, Richards BD, Jesse R, MacLean KA, Barrett FS, Cosimano MP, Klinedinst MA. Psilocybin-occasioned mystical-type experience in combination with meditation and other spiritual practices produces enduring positive changes in psychological functioning and in trait measures of prosocial attitudes and behaviors. J Psychopharmacol. 2018 Jan;32(1):49-69. doi: 10.1177/0269881117731279. Epub 2017 Oct 11. PMID 29020861
- See also: Study Website — http://www.bpru.org/spiritual-practice